CLINICAL TRIAL: NCT04966650
Title: Effectiveness of a Brief Nursing Advice in Promoting the Psychological Well-Being for University Students With Mild to Moderate Depressive Symptoms: A Randomized Controlled Trial
Brief Title: Brief Nursing Advice for University Students With Depressive Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: NTEC-2021-0379
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: The data collector is blinded. Those who analyses the data, using the electronic form, do not know the group belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): For the intervention group, participants will receive a 5-mins brief nursing advice incorporating with Social Cognitive Theory (SCT). The protocol is about the relationship between exercise and mental health, the advantages of increase physical activity and regular exercise, and highlight the consequence if not deal with the depressive symptoms. At the 2nd month, participants will be assessed their depression symptoms via questionnaire, followed up their progress of physical activity changes and given a booster intervention. At 6th months, subjects will be assessed their depression symptoms and the level of physical activity changes via questionnaire.
  Interventions: Behavioral: 5-mins brief nursing advice incorporating with Social Cognitive Theory (SCT)
- Control Group (No Intervention): A wellbeing leaflet from CHP will be provided to each participant. At the 2nd month, subjects will be assessed their depression symptoms via questionnaire, followed up their progress of physical activity changes and given another wellbeing leaflets. At 6th months, subjects will be assessed their depression symptoms the level of physical activity changes via questionnaire.

INTERVENTIONS:
Behavioral: 5-mins brief nursing advice incorporating with Social Cognitive Theory (SCT) — The protocol is about the relationship between exercise and mental health, the advantages of increase physical activity and regular exercise, and highlight the consequence if not deal with the depressive symptoms.
  Arms: Intervention group

SUMMARY:
1. Project title Effectiveness of a Brief Nursing Advice in Promoting the Psychological Well-Being for University Students with Mild to Moderate Depressive Symptoms: A Randomized Controlled Trial
2. Investigators Principal Investigator Ms. Tiffany PY CHAN, Doctor of Nursing (Year 3 candidate), School of Nursing, The University of Hong Kong (HKU) Nursing Officer, University Health Service, The Chinese University of Hong Kong (CUHK)

   Co-investigator Dr. William HC LI, Associate Professor, School of Nursing, The University of Hong Kong (HKU) Dr. Scotty Luk, Director, University Health Service, The Chinese University of Hong Kong (CUHK)
3. Study site Recruitment of participants will be conducted on campus in CUHK
4. Aims of the project This study aims to assess the effectiveness of a brief nursing advice in reducing depressive symptoms among university students who presented mild to moderate depressive symptoms at the University Health Service.
5. Outcomes The primary outcome of this study is the university students' decreasing level of depressive symptoms.

DETAILED DESCRIPTION:
University Students with Mild to Moderate Depressive symptoms University students experience a range of unique psychosocial stressors that increase their risk of major depression that are substantially higher than those found in the general population (Nahla, et.al., 2013). The prevalence rates of moderate to extremely severe depression symptom was 69.5% in Bangladesh (Islam, et.al., 2020), and 57.6% of the students suffered from moderate to extremely severe depression symptom among final-year medical students in India (Kumar, et.al.,2019), and a study showed that the prevalence of depression is particularly high among Australian university students (Farrer, et. al.,2016).

A report from the CHP in Hong Kong showed that the prevalence of mild to moderate, and severe depressive symptoms in adolescents and children were 51.1%, and 4.2% respectively in 2012 (CHP, 2020). However, a cross-sectional study of Hong Kong showed that a high proportion of the university students displayed depressive symptoms with 68.5% of them presented mild and moderate depressive symptoms, and 9% presented moderately severe to severe depressive symptoms (Lun, et. al., 2018). The result was higher than a similar survey (20.9%) conducted by the University of Hong Kong 10 years ago (Wong, et. al., 2006). Although almost 3 in every 5 undergraduate students (59.5%) in Hong Kong are likely to experience mild to moderate depressive symptoms, inadequate attention has been given in primary health care.

Health impact with Mild to Moderate Depressive symptoms Mild depression usually affects our daily activities and causes detectable symptoms in university students, and it is common but often remain unrecognized and treated inadequately (Klein, et. al., 2016). If the investigator can accurately diagnose depression when it is mild, and treating it effectively at this stage that can prevent the condition from worsening to become moderate or severe. The majority of suicide cases are linked with mental disorders, and most of them are triggered by severe depression. Suicide was the second leading cause of death among 15-29 year olds globally in 2015 (WHO, 2017). In Hong Kong, the number of suicides in the age-group 15 to 24 years increased in subsequent years from 54 in 2014, to 68 in 2015 and 75 in 2016 (DH, 2018).

Insufficient student mental health services within the University Campus In Hong Kong, only 3 out of 8 universities providing health services on campus. At the beginning of school term, students will be arranged to fill the mental wellness questionnaire from Office of Student Affairs, and they will be referred to see counselors or consult the doctor in school clinic if necessary. Only one university provides in-house psychiatric service, the student will be referred to In-house psychiatric service by OPD doctors. Other universities may refer to outside psychiatric service, with a long waiting queue for more than 6 months in Hospital Authority, or to receive private psychiatrist subsidized by university itself. For the current psychiatric service in one of the universities in Hong Kong, there is a total of 803 attendances (148 students) in 2018/19, with 5.4 visits per student, 79 of students have depression (53%), 55 students who had suicidal idea, plan or act (37%). A considerable increase in the demand for psychiatric services followed by an increase number of university students reported depressive symptoms (64 students in 2017-18 vs 79 students in 2018-19), consequently increased the waiting time for the consultation. Apart from the existing psychiatric consultation for those who presented severe depressive symptoms, there is an imperative need to develop and evaluate effective prevention strategies to help those university students with mild to moderate depressive symptoms.

Brief nursing advice for University Students with Mild to Moderate Depressive symptoms Evidence shows that a brief nursing advice is more feasible and cost-effective (Vijay, G.C.,et. al., 2015), and all very brief interventions for physical activity were acceptable and low cost. (Pears et. Al., 2015). It can increase physical activity in the short term when compared with usual care or more intensive interventions. Comparing to other interventions, such as cognitive behaviour therapy, which probably takes many weeks to implement but with only short-term effect in reducing depression (Stallman, et al.,2016). All nursing staff are well trained to provide a brief advice on mental health and thus no extra training is required. The intervention is suggested to deliver in a single session of no more than 5 min, that could be delivered in health checks or similar consultations (Vijay, G.C.,et. al., 2015). Students can receive brief nursing advice at the clinic.

Furthermore, nurses play as an important role in multidisciplinary collaboration in the University campus, such as Office of Student Affairs, faculty and department. They can refer their students to university clinic if the student is in needed. All urgent cases can be arranged to consult in-house psychiatrists within the same day.

If brief nursing advice in the campus can lower the depression symptoms of the university students, it can align with Department of Health in strengthening the primary health care and reduce the burden of tertiary healthcare. Due to the convenient location on campus, the intervention will be more accessible.

Why Physical activity? In general, the counselors or psychiatrists will focus on the stressors, or signs and symptoms of the university students which cause depression symptoms in the consultation visit. However, the evidence supporting physical activity as a treatment for mild-to-moderate depression, which is extensive and relatively uncontested. A precious study showed that university students who did exercise regularly reported fewer depressive symptoms than those who did not perform regular exercise (Lun, et. al., 2018). A study reported that both motivational and volitional elements are important in any intervention to increase physical activity in people with mild-to-moderate depression (Katarzyna, et. al., 2018). Physical activity was negatively related to the level of depression by severity among Undergraduate Students in Malaysia (Wan, et. al., 2020). Students with regular exercise towards the future experienced fewer depressive symptoms (Lun, et. al., 2018).

Theoretical or conceptual framework of how physical activity can help people reduce the depressive symptoms Theory-based interventions are more effective in changing behaviour than interventions that do not use a theoretical approach (Prestwich, A., et. al, 2014), and Social Cognitive Theory (SCT) is one of the most widely used theories in health behaviour research. SCT has guided the development of numerous physical activity interventions and its constructs are strongly associated with physical activity.

Research gap School-based intervention on mental health is found to be insufficient in both local and global university settings, and rarely discussed or reported in the literature. Besides, no study describe the theoretical or conceptual framework of brief intervention in health advice. The investigator hypothesized that brief nursing advice is effective to lower the severity of depressive symptoms of the university students with mild to moderate depressive symptoms.

7A. Study design: i. Study design We will conduct a Randomised Control Trial, with two-group pre-test and repeated post-tests, and a between-subjects design following CONSORT guideline. PHQ-9 questionnaires (PHQ-9) will be completed by the participants before and after receiving the intervention. The participants will be assessed their depression symptoms via questionnaire, followed up their progress of physical activity changes and given a booster intervention at 2nd month. At 6th month, participants will be assessed their depression symptoms via questionnaire. For the control group, participants will be given a health education leaflet and assessed their depression symptoms via questionnaire, followed up their progress of physical activity changes at 2nd month and 6th month. The researchers strictly adhere to the declaration of Helsinki.

ii. Settings The setting will be in University Health Service, CUHK campus.

iii. Subjects For the enrolment, all students who visit clinic will be assessed for the eligibility to join the study. The inclusion criteria include aged 18 aged or above, able to speak and read in Chinese, had presented mild to moderate depressive symptoms as identified by a minimum score of 5 on the Patient Health Questionnaire (PHQ-9), and will have at least 1 more year's study period in the university. The investigator will exclude those with actively suicidal, PHQ score >15-19 moderately severe, 20-27 severe depressive symptoms, or those who are receiving antidepressant medication or mental health service such as counselling or psychiatric consultation, or Athletes/ >150 minutes of moderate-intensity aerobic physical activity throughout the week, or at least 75 minutes of vigorous-intensity physical activity. For those are excluded in the study, all cases will be referred by medical doctors or in-house psychiatrists for follow up within the same day.

iv. Procedures

Randomization and allocation concealment Informed consent will be sought from each participant. The investigator will conduct baseline assessment, and randomization to allocate the subjects into intervention or control group. All procedure will be implemented in single room to ensure the privacy and to minimize the possibility of contamination.

Intervention group For the intervention group, participants will receive a 5-mins brief nursing advice incorporating with Social Cognitive Theory (SCT). The protocol is about the relationship between exercise and mental health, the advantages of increase physical activity and regular exercise, and highlight the consequence if not deal with the depressive symptoms. At the 2nd month, participants will be assessed their depression symptoms via questionnaire, followed up their progress of physical activity changes and given a booster intervention. At 6th months, subjects will be assessed their depression symptoms and the level of physical activity changes via questionnaire.

Control Group A wellbeing leaflet from CHP will be provided to each participant. At the 2nd month, subjects will be assessed their depression symptoms via questionnaire, followed up their progress of physical activity changes and given another wellbeing leaflets. At 6th months, subjects will be assessed their depression symptoms the level of physical activity changes via questionnaire.

After the completion, the subject will be received a $50 cash coupon for the incentive.

v. Data analysis All data will be entered and analyzed by using SPSS for Window, v. 26. Independent t-test will be used to compare the change in depressive symptoms before and after intervention between the two groups. The investigator will use the 9-item Patient Health Questionnaire (PHQ-9) for the measurement tool. It is a valid and reliable tool for assessing depressive symptoms in Hong Kong general population. It is used to monitor the severity of depression and response to treatment.

vi. Timeline Research procedure Month/ Year 2021-2022 Aug Sep Oct Nov Dec Jan Feb Mar Apr May Jun Preparation of questionnaire and recruitment Recruitment and data collection 2nd month post-intervention evaluation 6th month post-intervention evaluation Data management, analysis, and report writing

8. Drug investigation: Nil 9. Describe any unusual or discomforting procedures to be used: Nil. 10. Are there any hazards associated with the investigation? No 11. Direct access to source data/documents The raw data will be stored in the USB and locked in a safe cabinet by the Principal Investigator. Only the Investigator will be permitted to access to raw data or study record. The data will be kept for 3 years after the study completed.

12. Dissemination of study result The research findings will be presented in collective form in local and international conferences and published in international peer reviewed journals.

13. Consent Eligible participants will be invited to participate in the study by giving a written consent.

14. Conflict of interest: None 15. Financing and insurance: None

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria include aged 18 aged or above, able to speak and read in Chinese, had presented mild to moderate depressive symptoms as identified by a minimum score of 5 on the Patient Health Questionnaire (PHQ-9), and will have at least 1 more year's study period in the university.

Exclusion Criteria:

* We will exclude those with actively suicidal, PHQ score >15-19 moderately severe, 20-27 severe depressive symptoms, or those who are receiving antidepressant medication or mental health service such as counselling or psychiatric consultation, or Athletes/ >150 minutes of moderate-intensity aerobic physical activity throughout the week, or at least 75 minutes of vigorous-intensity physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
depression symptoms | o month, 2nd month, 6 month
  Change of the level of depression symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung Li, Study Director — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibrahim AK, Kelly SJ, Adams CE, Glazebrook C. A systematic review of studies of depression prevalence in university students. J Psychiatr Res. 2013 Mar;47(3):391-400. doi: 10.1016/j.jpsychires.2012.11.015. Epub 2012 Dec 20. PMID 23260171